CLINICAL TRIAL: NCT00476515
Title: Multicenter Trial Using Multi-dose Rituximab as Induction and Desensitization Therapy for Patients on the Waiting List for Kidney Transplant With a Positive Donor Specific Crossmatch to a Living Donor
Brief Title: Rituximab Therapy for Patients on Kidney Transplant Waiting List With Positive Donor Specific Crossmatch to Living Donor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol to be revised
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Biogen (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nina Tolkoff-Rubin, MD, Physician, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006P002059
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Kidney Insufficiency
Keywords: Kidney transplantation; Donor specific antibodies; Positive cross match
MeSH Terms: conditions — Renal Insufficiency | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): this study has only one arm as treatment group.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — the recommended dosage of Rituximab is 375 mg/m2 given as an IV infusion once weekly for four doses (days 1, 8, 15, and 22).
  Other Names: Rituxan

SUMMARY:
Primary Objectives:

* Conversion of a positive donor specific cross-match to a living donor to a negative cross-match thereby allowing successful renal transplantation.
* Transplant success or failure following the desensitization protocol.
* Determination of the effect of rituximab on the kinetics of donor specific antibodies (DSA).
* Determination of the effect of rituximab on the kinetics of B-cell subpopulations in peripheral blood and/or secondary lymphoid organs (lymph node biopsies at time of transplant, if available) in both responders and non-responders using flow cytometry and/or immunohistochemistry.

Secondary Objectives:

-Decrease in incidence of humoral rejection to less than 50 % at 1 year.

DETAILED DESCRIPTION:
For patients with a donor specific antibody, a protocol of plasmapheresis and intravenous immunoglobulin has been used to remove circulating antibodies and suppress antibody production. While this therapy is effective at enabling transplantation, it has a reported failure rate of 50% (Personal communication, Johns Hopkins' group); it is expensive (average cost of protocol $55,000.00 does not include transplant surgery costs; personal communication: Johns Hopkins' group) and may be fraught with infectious complications particularly when combined with current immunosuppression protocols.

To date, there is no effective treatment protocol designed to desensitize end stage renal disease patients with a high Panel of Reactive Antibodies (PRA) (i.e., >70%). Patients with elevated PRA levels have a longer median organ waiting time when compared to those with lower PRA. Patients with elevated PRA have decreased allograft survival when compared to controls. It has been reported that 50% of cadaveric kidneys transplanted into high PRA recipients (>20%) suffered of rejection within 6 months of transplantation.

Pathophysiologically, an elevated PRA or a donor specific antibody is acquired through the sensitization of the host against major histocompatibility antigens (HLA) following multiple blood transfusions, prior pregnancy or organ transplantation. The constant levels of anti-HLA antibodies are maintained through the persistent stimulation of naïve and memory B-cells by these antigens. The number of patients with a high PRA and/or donor specific antibodies is expected to increase as more patients with failed kidney transplants are entering the waiting list.

Although initially introduced for the treatment of neoplasms, the humoral immunosuppressant effects of Rituximab have been shown to have clinical significance. In an attempt to understand the humoral immunosuppressant effects of Rituximab Gonzalez-Stawinski et al., reported the effects of the monoclonal on a de-novo and memory humoral immune response. Their work showed that Rituximab interferes with both primary and secondary humoral responses by eliminating B-cells prior to antigen exposure thus interfering with differentiation into antibody secreting cells and specific antibody production (Gonzalez-Stawinski)

Enthusiasm for these data resulted in small, single center experiences using Rituximab in the post-transplant and pre-transplant settings. Post-transplantation, Becker et al. utilized Rituximab as rescue therapy in 4 kidney transplant patients who developed acute humoral rejection. These patients had failed conventional rescue therapy (high dose intravenous steroids, and plasmapheresis with IVIg), but transplants were salvaged by a single dose of Rituximab (375mg/M2) as demonstrated by improvements in creatinine clearances. Also in a post-transplant setting, Samaniego et al. successfully utilized Rituximab in a small population of highly sensitized renal transplant patients with positive donor specific crossmatch who failed the standard plasmapheresis and IVIg protocol. Pre-transplantation, Vieira et al were able to reduce the concentrations of anti-HLA antibodies after the administration of a single dose of Rituximab. Fifty percent of these patients had their PRA's decrease by nearly 40% of baseline.

In these small clinical reports, Rituximab has been an effective humoral immunosuppressant that eliminates the cell population responsible for anti-HLA antibody production by virtue of the modulation of naïve or memory B-cells prior to/or during HLA stimulation. However, the effect of a schema of multiple doses of Rituximab on donor specific crossmatch is yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Active status on a kidney transplant waiting list for over 2 years
* Donor specific antibody titer <= 1:128 (Class I, Class II or both) by cytotoxicity
* Signed and dated informed consent
* Age ≥ 18 years
* Positive cross-match against a living donor

Exclusion Criteria:

* Donor specific antibody titer greater than 1:128 (Class I, Class II or both) by cytotoxicity
* Inactive status on a kidney transplant list
* Treatment with any investigational agent within 4 weeks of screening or 5-half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera/Rituxan)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Positive history of HIV
* Positive history of Hepatitis B and/or Hepatitis C
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum or urine pregnancy test should be performed for all women of childbearing potential within 7 days of treatment)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of psychiatric disorder
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Laboratory Exclusion Criteria (at Screening)
* Hemoglobin: < 7g/dL
* Platelets: <100,000/mm3
* AST or ALT >2X Upper limit of normal
* Known history of positive Hepatitis B or C serology
* Immunization status to be confirmed per transplant protocol. Review of the subject's immunization status for the following vaccinations will be ascertained: tetanus; diptheria; influenza; pneumococcal polysaccharide; Varicella; measles, mumps and rubella (MMR); and hepatitis B. Subjects who are considered to be at high risk for hepatitis B virus (HBV) infection and for whom the investigator has determined that immunization is indicated should complete the entire HBV vaccine series (per routine dialysis protocol) at least 4 weeks prior to participation in the study.

Immunization with a live vaccine is specifically excluded during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Subjects who convert to a negative donor specific crossmatch or eliminate donor specific antibody will be considered a TREATMENT SUCCESS and will undergo target living donor transplantation in 3-5 days | 4 weeks after the final dose of Rituximab

CONTACTS AND LOCATIONS:
Overall Officials: Nina Tolkoff-Rubin, MD, Principal Investigator — Massachusetts General Hospital